CLINICAL TRIAL: NCT01034514
Title: 4D-CT-based Ventilation Imaging for Adaptive Functional Guidance in Radiotherapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Billy W. Loo Jr. (Other)
Responsible Party: Sponsor-Investigator, Billy W. Loo Jr., Associate Professor of Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUN0034; SU-04232009-2382 (Other: Stanford University)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Positron-Emission Tomography; Tomography, Emission-Computed, Single-Photon; Pentetic Acid; Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 4DCT arm (Experimental): Patients breathe in 99mTc-DTPA and then undergo ventilation scans using a SPECT scanner over 2 hours. Patients also receive 99mTc-MAA IV and then undergo perfusion scans using a SPECT scanner over 2 hours. Patients may also undergo a pre- and post-treatment Xe-CT ventilation scan over 15 minutes and a pre-treatment 4D-CT scan over 5-10 minutes.
  Interventions: Device: Real-time Position Management system; Device: Discovery ST multislice PET/CT scanner; Device: Infinia Hawkeye SPECT/CT gamma camera; Device: Pinnacle3 treatment planning system; Device: SKYLight nuclear camera; Drug: DTPA; Drug: TECHNETIUM TC 99M MAA

INTERVENTIONS:
Device: Real-time Position Management system — Standard of Care
  Other Names: RPM System
Device: Discovery ST multislice PET/CT scanner — Standard of Care
  Other Names: Positron Emission Tomography
Device: Infinia Hawkeye SPECT/CT gamma camera — Standard of Care
  Other Names: Single-photon emission computed tomography
Device: Pinnacle3 treatment planning system — Standard of Care
  Other Names: Radiation Treatment Planning
Device: SKYLight nuclear camera — Standard of Care
  Other Names: Philips Medical Systems
Drug: DTPA — 1 mCi; inhalation
  Other Names: DRAXIS Specialty Pharmaceuticals Inc.
Drug: TECHNETIUM TC 99M MAA — 3 mCi; iv
  Other Names: DRAXIS Specialty Pharmaceuticals Inc.

SUMMARY:
To develop and investigate a novel radiotherapy technique for preserving lung function based on a map of lung function.

ELIGIBILITY:
Inclusion Criteria:

* Eligible disease(s)/stage(s) AJCC Stage I, II, III or IV lung cancer of any histology to be treated using radiotherapy will be eligible for this study. Note that we will carefully consider the inclusion of cases with turbulent flow or greater flow velocities (Cabahug et al., 1996; Crawford et al., 1990) and COPD cases (Magnant et al., 2006) due to the impaction of aerosol particles in central airways.
* Allowable type and amount of prior therapy. Any types and amounts of prior therapy will be allowed for this study.
* Age restriction and/or gender/ethnic restrictions
* Patients must be greater than or equal to 18 years of age.
* There are no gender or ethnic restrictions.
* Life expectancy restrictions - None.
* ECOG or Karnofsky Performance Status
* Not employed. Note that patients will need to be sufficiently healthy to undergo audiovisual (AV) biofeedback to generate high quality 4D-CT images.
* Requirements for organ and marrow function None.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Children (less than 18 years of age), pregnant women, Stanford employees or students, or prisoners will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-06-24 (Actual)

PRIMARY OUTCOMES:
The overall correlation between the 4D-CT and the SPECT ventilation images. | 24 months

SECONDARY OUTCOMES:
The difference between the local ventilation at simulation and during the treatment. Dose-volume or functional dose-volume metrics. The regression coefficient between the regional ventilation and time. The mean dose to the high-functional lung region. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Billy Loo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States